CLINICAL TRIAL: NCT06564155
Title: Inturlekin 33 in Ankylosing Spondylitis Patients and Its Relationship to Subclinical Atherosclerosis
Brief Title: Inturlekin L33 in Ankylosing Spondylities Patients and Its Relation to Subclinical Atherosclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Hussein AbuAli, Principial investigator, Assiut University
Other Study IDs: IL33 in Ankylosing spondylites
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: None Retained — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ankylosing spondylities patients: detect level of IL33 in serum of AS patients
  measure carotid intima media thickness by caroid dupex
  Interventions: Device: carotid duplex
- control persons: detect level of IL33 in serum of normal control group
  measure carotid intima media thickness by caroid dupex
  Interventions: Device: carotid duplex

INTERVENTIONS:
Device: carotid duplex — measure Carotid intima media thickness

SUMMARY:
detect level of Inturlekin 33 in ankylosing spondyilits patient

measure CIMT (carotid intima media thickness ) by carotid duplex to detect subclinical atherosclerosis in ankylosing spondyitis patients

detect the relation between IL33 and subclinical atherosclerosis in Ankylosinig Spondylitis patients

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS), a type of SpA, is an autoimmune disease that mainly involves, sacroiliac joints (SIJs) and their adjacent soft tissues, such as tendons and ligaments. The main clinical manifestations include back pain and progressive spinal rigidity as well as inflammation of the hips, shoulders, peripheral joints and fingers/toes. In addition, there are extra-articular manifestations.

Cardiovascular disease has become the first cause of death for patients with ankylosing spondylitis (AS).

Patients with ankylosing spondylitis (AS) have an increased cardiovascular morbidity and mortality . Accelerated atherosclerosis caused by a systemic inflammatory response has been reported to be an important risk factor for increased cardiovascular risk for autoimmune diseases.

Interleukin (IL)-33 is a cytokine belonging to the IL-1 family and was recently identified as a ligand for ST2, .the serum levels of IL-33/sST2 were remarkably higher in the patients with AS than the healthy groups .

Pervious studies confirm the importance of IL-33/ST2 axis in the process of atherosclerosis, and indicate its ambiguous function in immune response, whether as proinflammatory cytokine in advanced atherosclerotic lesions, or as profibrotic, in early lesions.

Previous study shows increased CIMT in AS patients without traditional cardiovascular risk factors compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed as Ankylosing Spondylitis
* Age (20-40)

Exclusion Criteria:

* Patients with other rheumatic diseases/other SPA types

  * Participants with history of CVD event in past or present
  * Patient experiencing cardiovascular revascularization surgery or cerebrovascular disorder within past 6 months.
  * Patient with other risk factor for atherosclerosis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * patient diagnosed as Ankylosing Spondylitis according to ASAS 2009
  * Age (20-40)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
detect level of IL33 in AS patients | 3 years
  measure level of IL33 in the serum of AS patients measure caroid intima media thickness CIMT in AS patients

SECONDARY OUTCOMES:
detect the reation between IL33 and subclinical atherosclerosis in AS patients | 3 years
  measure caroid intima media thickness CIMT in AS patients

REFERENCES:
- [Result] Li GX, Wang S, Duan ZH, Zeng Z, Pan FM. Serum levels of IL-33 and its receptor ST2 are elevated in patients with ankylosing spondylitis. Scand J Rheumatol. 2013;42(3):226-31. doi: 10.3109/03009742.2012.735700. Epub 2013 Feb 15. PMID 23409750